CLINICAL TRIAL: NCT06987643
Title: A Double-Blind, Placebo-Controlled, Proof-of-Concept Clinical Study of the P38 Alpha Kinase Inhibitor Neflamapimod on Recovery After Moderate to Severe Acute Ischaemic Stroke
Brief Title: A Clinical Study to Investigate the Effect of Oral Neflamapimod on Motor Recovery After Acute Ischaemic Stroke
Acronym: RESTORE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: EIP Pharma Inc (Industry)
Collaborators: CervoMed, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRVO24-NFD-601
Record Dates: First submitted 2025-05-05; First posted 2025-05-23 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Moderate to Severe Acute Ischaemic Stroke; Ischaemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — VX-745

STUDY DESIGN:
Intervention Model Description: This is a double-blind, randomised, parallel arm, placebo-controlled, multicentre, Phase 2b exploratory study of neflamapimod in participants with moderate to severe acute ischaemic stroke. Participants enrolled into cohort 1 are randomized 1:1 (neflamapimod:placebo), dosing 3 times per day. Participants enrolled into cohort 2 are randomized 1:1 (neflamapimod:placebo), dosing 2 times per day.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cohort 1 neflamapimod (Active Comparator): Neflamapimod will be administered with food for 12 weeks in subjects with Moderate to Severe Acute Ischaemic Stroke. Subjects will receive 3 capsules per day (TID) with food (i.e., with the morning, mid-day and evening meals).
  Interventions: Drug: Neflamapimod
- Cohort 1 placebo (Placebo Comparator): Placebo will be administered with food for 12 weeks in subjects with Moderate to Severe Acute Ischaemic Stroke. Subjects will receive 3 capsules per day (TID) with food (i.e., with the morning, mid-day and evening meals).
  Interventions: Drug: Placebo
- Cohort 2 placebo (Placebo Comparator): Placebo will be administered with food for 12 weeks in subjects with Moderate to Severe Acute Ischaemic Stroke. Subjects will receive 2 capsules twice per day (BID) with food (i.e., with the morning and evening meals).
  Interventions: Drug: Placebo
- Cohort 2 neflamapimod (Active Comparator): Neflamapimod will be administered with food for 12 weeks in subjects with Moderate to Severe Acute Ischaemic Stroke. Subjects will receive 2 capsules twice per day (BID) with food (i.e., with the morning and evening meals).
  Interventions: Drug: Neflamapimod

INTERVENTIONS:
Drug: Neflamapimod — Neflamapimod is a highly specific inhibitor of the intra-cellular enzyme mitogen-activated protein kinase14 (p38α) provided in 40mg capsules
  Other Names: VX-745
  Arms: Cohort 1 neflamapimod; Cohort 2 neflamapimod
Drug: Placebo — Placebo is a capsule that looks just like neflamapimod but without the active ingredients
  Arms: Cohort 1 placebo; Cohort 2 placebo

SUMMARY:
The purpose of this interventional study is to determine whether neflamapimod can improve residual physical disability and/or cognitive dysfunction after Moderate to Severe Acute Ischaemic Stroke.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants must be aged 45 years or over at the time of signing the informed consent.
* Confirmed acute ischaemic stroke in the anterior circulation (middle or anterior cerebral artery) with onset of symptoms between 2 and 7 days prior to screening and evaluation.
* National Institutes of Health Stroke Scale (NIHSS) score between 5 and 20 (inclusive) and exhibiting unilateral motor deficit (i.e. motor NIHSS ≥ 2 on affected side of the body).
* Fugl-Meyer Assessment of Motor Recovery after Ischaemic Stroke (FMMS) total motor components score of 80 or below.
* No history of learning difficulties that may interfere with their ability to complete the cognitive tests.

Exclusion Criteria:

* Evidence of progressive or unstable stroke or intra-cerebral haemorrhage in the opinion of the investigator
* Participants needing carotid surgery within 3 months
* Ongoing major and active psychiatric disorder and/or other concurrent medical condition that, in the opinion of the Investigator, might compromise safety and/or compliance with study requirements.
* History of alcohol or drug abuse within the previous 2 years.
* Poorly controlled clinically significant medical illness, such as hypertension (blood pressure >180 mmHg systolic or 100 mmHg diastolic); myocardial infarction within 6 months; uncompensated congestive heart failure or other significant cardiovascular, pulmonary, renal, liver, infectious disease, immune disorder, or metabolic/endocrine disorders or other disease that would interfere with assessment of drug safety in the opinion of the Investigator.
* Abnormal laboratory tests that, in the Investigator's assessment, mean that a participant is not appropriate for participation in this study, including, but not limited to:

  1. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2.0

     × the upper limit of normal (ULN),
  2. Total bilirubin >1.5 × ULN, and/or
  3. International Normalised Ratio (INR) >1.5 NOTE: Participants with Gilbert's syndrome can be included with total bilirubin >1.5 x ULN as long as direct bilirubin is ≤ 1.5 x ULN)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-28 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to Week 12 in Fugl-Meyer Assessment of Motor Recovery after Stroke (FMMS) motor score (upper and lower) and total score | From enrollment until the end of treatment at 12 weeks
  The FMMS test has a maximum upper motor score of 66, maximum lower motor score of 34, and a maximum total score of 212, where an increase indicates improved motor function while a decrease indicates worsening impairment.
Change from baseline to Week 12 in the Timed Up and Go Test (TUG) | From enrollment until the end of treatment at 12 weeks
  The TUG test is recorded in seconds. The test has no minimum or maximum value, and an increase in the time required to complete the TUG is a worse outcome.
Change from baseline to Week 12 in National Institutes of Health Stroke Scale (NIHSS) motor score | From enrollment until the end of treatment at 12 weeks
  Scores for the NIHSS range from 0 to 42 where higher scores indicate greater impairment/worsening.

SECONDARY OUTCOMES:
Proportion of participants with Modified Rankin Scale (mRS) score of ≤ 2 at Week 12 | From enrollment until the end of treatment at 12 weeks
  The mRS scores range from 0 (no symptoms) to 6 (death) where higher scores indicate greater impairment/worsening.
Change from baseline to Week 12 in mean Barthel score | From enrollment until the end of treatment at 12 weeks
  The Barthel Index (BI) for Activities of Daily Living scores range from 0 (total dependency) to 100 (independent) where higher scores indicate greater independence/improvement.

CONTACTS AND LOCATIONS:
Locations (12):
- Australia (12):
  - Campbelltown Hospital, Campbelltown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Western Health- Sunshine Hospital, St Albans, Victoria

IPD SHARING:
Plan to Share IPD: No